CLINICAL TRIAL: NCT00337376
Title: A Phase I Study of the mTOR Inhibitor Rapamycin (Rapamune, Sirolimus) in Combination With Abraxane (Paclitaxel Protein-bound Particles) in Advanced Solid Cancers
Brief Title: A Study of the mTOR Inhibitor Rapamycin (Rapamune, Sirolimus) in Combination With Abraxane in Advanced Solid Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Maysa Abu-Khalaf, Principal Investigator, Yale University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0511000860
Record Dates: First submitted 2006-06-13; First posted 2006-06-15 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2014-01

CONDITIONS: Advanced Solid Cancers
MeSH Terms: interventions — Sirolimus; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Rapamune; Drug: Abraxane

INTERVENTIONS:
Drug: Rapamune — Dose escalation as follows: 5mg PO, 10mg PO, 20mg PO, 40mg PO
  Other Names: Rapamycin; Sirolimus
Drug: Abraxane — intravenous administration of 100mg/m2 Abraxane over 30 minutes, weekly for three out of four consecutive weeks.
  Other Names: Albumin-bound paclitaxel

SUMMARY:
Rapamycin is a drug that has been approved by the Food and Drug Administration (government) for use in patients receiving a kidney transplant to prevent the patient's body from rejecting the transplanted kidney. It has shown antitumor effects in the laboratory, but has not been approved at this time for the treatment of cancer. Abraxane is a new form of chemotherapy that has been approved by the Food and Drug Administration for the treatment of metastatic breast cancer, and is a promising drug that is being evaluated in clinical trials for treatment of other cancers. This is a phase I study designed to find out if different doses of Rapamycin, when combined with Abraxane, are safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-confirmed advanced solid tumors.
* For patients with metastatic breast cancer, there will be no restriction on prior therapy. For patients with other advanced solid tumors, they must be refractory to standard therapy or for which no curative standard therapy exists, to be considered. Metastatic disease, if present, should not be progressing so as to require palliative treatment within 4 weeks of enrollment based on clinical assessment by the investigator.
* Development of new lesions or an increase in preexisting lesions on bone scintigraphy, CT, MRI or by physical examination. Patients in whom the sole criterion for progression is an increase in a biochemical marker, e.g., carcinoembryonic antigen (CEA), or an increase in symptoms, are not eligible.
* No radiotherapy, treatment with cytotoxic agents, or treatment with biologic agents within the 4 weeks prior to beginning treatment on this study (6 weeks for mitomycin or nitrosoureas). At least 2 weeks must have elapsed from any prior surgery or hormonal therapy. Patients must have fully recovered from the acute toxicities of any prior treatment with cytotoxic drugs, radiotherapy or other anti-cancer modalities (returned to baseline status as noted before most recent treatment). Patients with persisting, stable chronic toxicities from prior treatment ≤ grade 1 are eligible.
* Age ≥18 years.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A).
* Life expectancy of greater than 3 months.
* Patients must have normal organ and marrow function as defined below:

Hemoglobin ≥ 9 g/dL leukocytes ≥3,000/mcL absolute neutrophil count ≥1,500/mcL platelets ≥100,000/mcL total bilirubin within normal institutional limits AST(SGOT)/ALT(SGPT)2.5 X institutional upper limit of normal creatinine within 1.5 x ULN OR creatinine clearance ≥50 mL/min/1.73 m² for patients with creatinine levels ≥1.5 ULN.

* Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and must have a negative serum or urine pregnancy test within 1 week prior to beginning treatment on this trial. Pregnant and nursing patients are excluded because the effects of the combination of Abraxane and Rapamycin on a fetus or nursing child are unknown. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. Sexually active men must also use appropriate contraception method and should not father a child while receiving therapy during this study.
* Ability to understand and the willingness to sign a written informed consent document.
* Fasting serum cholesterol <350 mg/d L and triglycerides < 400 mg/ d L.
* Biopsy is required but patients or physicians may opt out of this part of the trial if sufficient justification is provided. Justification must be provided to the PI in writing indicating excessive physical risk or psychological trauma if biopsy is taken

Exclusion Criteria:

* Patients must be 4 weeks from chemotherapy or radiotherapy and have recovered from any adverse events
* Patients may not be receiving any other investigational agents.
* Patients with known active brain metastases. Patients must have completed definitive treatment for brain metastases, at least 4 weeks prior to first dose on this study, and off steroids for at least 2 weeks, with stable or regressing CNS lesions by MRI or CT scan, and no evidence of new lesions.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in study.
* Peripheral neuropathy ≥ Grade 2
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because the investigational agents may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued if the mother is treated.
* HIV-positive patients are ineligible because these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy and the potential pharmacokinetic interaction between antiretroviral therapy and the investigational agents.
* All herbal and alternative medications should be discontinued while on study, these include but not limited to: Hydrastis canadensis (goldenseal), Uncaria tomentosa (cat's claw) Echinacea angustifolia
* Use of any of these medications within 1 week, prior to the first dose of treatment: cyclosporine, diltiazem, ketoconazole, rifampin, fluconazole, delavirdine, nicardipine, pioglitazone and sulfonamides, erythromycin, clarithromycin, itraconazole, metoclopramide, nevirapine, Phenobarbital, phenytoin, indinavir fosamprenavir, ritonavir, efavirenz, nefazadone, and St. John's wort.
* Consumption of grapefruit juice is prohibited during the study.
* Requirement for treatment with warfarin (Coumadin), immunosuppressive agents or chronic steroids
* Prior therapy with rapamycin, rapamycin analogs or experimental agents targeting mTOR
* Prior Abraxane therapy
* Active infection or treatment for systemic infections within 14 days of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To determine the safety, dose-limiting toxicities, and maximum tolerated dose of weekly oral Rapamycin in combination with weekly intravenous Abraxane for three out of four consecutive weeks in patients with advanced solid cancers. | upon completion of study

SECONDARY OUTCOMES:
to determine if weekly administration of Rapamycin changes the pharmacokinetic profile of weekly Abraxane | upon completion of study
To determine pre and post therapy changes in p70S6K in peripheral mononuclear cells in patients treated with oral Rapamycin and Abraxane | Upon completion of study
To evaluate changes in the phosphorylation of p70S6K on tumor tissue and to determine the correlation with phosphorylation of p70S6K in the peripheral mononuclear cells, in patients who give consent to pre and post tumor biopsies | upon completion of study

CONTACTS AND LOCATIONS:
Overall Officials: Maysa Abu-Khalaf, M.D., Principal Investigator — Yale University
Locations (1):
- Yale Comprehensive Cancer Center at Yale University School of Medicine, New Haven, Connecticut, United States